CLINICAL TRIAL: NCT05453760
Title: Lung Ultrasound in the Early Detection of Postoperative Pulmonary Complications After Esophagectomy: A Prospective Observational Study
Brief Title: Lung Ultrasound in the Early Detection of Postoperative Pulmonary Complications After Esophagectomy
Acronym: OESOLUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0076; 2022-A00655-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Neoplasm
Keywords: Thoracic Esophagectomy; Esophagectomy; Postoperative pulmonary complications; lung ultrasound; critical care
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The perioperative management of esophageal cancer has evolved considerably in recent years.

Over the last 30 years, postoperative mortality has been steadily decreasing. However, respiratory morbidity remains high (30-40%). This is due to the procedure itself requiring a thoracic approach and intraoperative unipulmonary ventilation. The postoperative pulmonary complications (PPCs) are multiple: bronchial congestion, atelectasis, pneumopathy, acute respiratory failure, liquid pleural effusion, pneumothorax.

In general, prevention and early treatment are aimed at limiting the evolution towards acute respiratory failure requiring ventilatory assistance.

Chest radiography is essential for the presumptive diagnosis of pneumopathy in particular, but the interpretation of the images may be difficult.

Thoracic computed tomography (CT) is the gold standard because it is sensitive and can discriminate among differential diagnoses. This is difficult to perform: it requires intra-hospital transport of patient, who is often in acute respiratory failure, and the availability of an examination area.

Lung ultrasound is used at the bedside for diagnosis of lung infection in intensive care unit. This has a sensitivity close to thoracic CT and has the advantage of being feasible at any time, does not require transport of the patient and is not irradiating.

Lung ultrasound allows early detection of the need for ventilatory support in postoperative major abdominal surgery . In addition, the sensitivity of lung ultrasound is close to that of CT, allowing this examination to be relied upon.

The main objective of the study is to determine the role of lung ultrasound (LUS) in the prediction of postoperative pulmonary complications within one hour after extubation. The secondary objectives are to determine the performance of lung and diaphragmatic ultrasound (DUS) on postoperative day 1 and to establish a predictive model integrating LUS, DUS, and clinical variables to improve early identification of patients at risk of postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic Esophagectomy

Exclusion Criteria:

* Emphysema Death during surgery Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort study of esophagectomy patients in a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the Lung ultrasound score | at Day 0 (within 1 hour of tracheal extubation)

SECONDARY OUTCOMES:
Area under the curve (AUC) of the Lung ultrasound score at Day 1 | Day 1
Diaphragmatic excursion is measured via subcostal diaphragmatic ultrasound performed during the patient's clinical examination | at Day 0, Day 1 and Day 3
The presence of condensations on pleuropulmonary ultrasound in the ICU | at Day 0, Day 1 and Day 3
The presence of pleural effusion at D0, D1 or D3 | at Day 0, Day 1 and Day 3
Complications according to the Dindo-Clavien classification | at Day 7
Mortality at D30 according to the LUS score at day 0 and day 1 | Between Day 0 et Day 30
Correlation between the LUS score on day 0 and day 1 and the mechanical energy delivered to the lung during surgery. | between the day 0 and the day 1
Assess whether diaphragmatic excursion measured on day 0, day 1, ans day 3 is predictive of CPPO within 7 days post-operatively. | Within 7 days post-operatively.
Evaluate whether the LUS score on day 1 correlates with PaO2/FiO2 on day 1. | A day 1.
Predictive model for postoperative pulmonary complications | At day 1
  Establish a predictive model integrating LUS, DUS and clinical variables (age, ASA score, surgical approach)

CONTACTS AND LOCATIONS:
Overall Officials: Cédric CIRENEI, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France